CLINICAL TRIAL: NCT01423383
Title: Epidemiology Study of Keloid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tirgan, Michael H., M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: Tirgan 11-04
Record Dates: First submitted 2011-08-23; First posted 2011-08-25 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Keloid
Keywords: Keloid
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Random Populations: The aim of this study is to determine the prevalence and incidence of keloid in large populations.

SUMMARY:
Although keloid is a very common condition; there are no statistics as to its true incidence and prevalence, neither in United States, nor elsewhere in the world. This trial intends to capture epidemiological data about this disease in a large population sample.

DETAILED DESCRIPTION:
The purpose of current trial is to establish a robust database of incidence and prevalence of keloid, as well as prevalence of familial keloid, in various ethnic groups. Study sample size is 100,000 random individuals who will fill out either a web survery or a paper questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Age above 18 to answer the survey questions
3. Parents shall respond on behalf of their minor children

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General population will be sampled randomly
Sampling Method: Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2011-09; Primary Completion 2020-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of various clinical findings will be determined at the end of Survey. | Two Years
  This will be a prospective online and paper based survey with an estimated 100,000 responders participating in two years. Statistics will be descriptive. The prevalence of various clinical findings will be determined at the end of Survey. Findings will be correlated with the source of the data, online, or paper questionnaire, as well as the locations where the paper questionnaires surveys were placed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Tirgan, MD, Study Chair — St. Luke's-Roosevelt Hospital Center
Locations (1):
- Michael H. Tirgan, MD, New York, New York, United States

REFERENCES:
- See also: This is the official website of this study. — http://www.EpidemiologyStudy.com